CLINICAL TRIAL: NCT03101215
Title: Workload of Water Polo Players Following a Phosphorus Manipulated High Carbohydrate Meal
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Omar Obeid, Professor, American University of Beirut Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: NUT:OO:24
Record Dates: First submitted 2017-03-24; First posted 2017-04-05 (Actual); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Energy Expenditure
MeSH Terms: interventions — Phosphorus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): glucose drink (100g) with placebo tablets
  Interventions: Dietary Supplement: phosphorus
- phosphorus (Active Comparator): Glucose drink (100g) with phosphorus tablets (400 mg of phosphorus)
  Interventions: Dietary Supplement: phosphorus

INTERVENTIONS:
Dietary Supplement: phosphorus — adding of phosphorus to high carbohydrate meal

SUMMARY:
Phosphorus is a widely used sport supplement. Most athletes who use it follow a phosphorus loading approach which consists of a weeklong phosphorus intake of 3-4 gr per day for optimal effect. The ergogenic potential of phosphorus is believed to be related to several factors including its ability to a) enhance ATP availability for energy expenditure and b) increase plasma content of 2.3-DPG (2.3-disphosphoglycerate) that is known to reduce oxygen affinity to hemoglobin and consequently enhances its release in the exercising tissue. Additionally, phosphorus was reported to increase peripheral glucose uptake and thus glycogenesis and glycogen storage. We have recently observed that the peripheral glucose uptake was stimulated by co-ingestion of phosphorus with meal, while pre ingestion failed to do so. Thus it is reasonable to postulate that phosphorus co-ingestion with meal improves ergogenesis through enhancing glycogen storage. The aim of this experiment is to investigate whether acute phosphate supplementation of a glucose load is responsible for the performance enhancement. This may help in explaining the controversies surrounding the impact of phosphorus on performance. A cross over study will be conducted on water polo players. In brief, overnight fasted subjects, will be given glucose load with or without phosphorus. Three hours later their performance will be measured using an ergometer cycling machine.

DETAILED DESCRIPTION:
The use of phosphorus as ergogenic aid has been widely reported and researched (Buck et al, 2013). Most of the research has centered on its chronic intake effect, usually for a loading period of 3-6 days (Kopec et al, 2015). The benefits of phosphate supplementation on athletic performance have been attributed to several potential factors, like increased maximal oxygen uptake and improved cardiac output (Folland et al, 2008). The underlying mechanisms were hypothesized to be the increased plasma content in 2.3-DPG (2.3-disphosphoglycerate) which may be a factor in reduced oxygen affinity to hemoglobin and consequent enhanced release in the exercising tissue (Di Caprio et al, 2015). Other lines of investigation, which were based on blood analysis and hypophosphatemia's effect on metabolism (Lichtman et al, 1971), and the rate of glycogenolysis in exercising muscle and rate of inorganic phosphorus (Chasiotis, 1988), attribute the beneficial effects of phosphate supplementation to higher extracellular concentration leading to increased ATP formation. A positive effect of phosphate supplementation was detected independently of 2.3-DPG in a recent study (Czuba et al, 2009). Additionally, increased phosphate availability was reported to increase peripheral glucose uptake (Khattab et al 2015) and stimulate glycogen synthesis (Xie et al, 2000). The failure of acute phosphate supplementation alone, without carbohydrate, to affect athletic performance (Galloway et al, 1996) may be partially attributed to low glycogen availability. We hypothesize that phosphorus exerts its effect acutely through increasing glycogen content of liver and muscles. Hence the acute effect of Phosphorus in physiologic doses on athletic performance may reveal another aspect of phosphate supplementation. If an improvement in work output is detected, as a significant difference in Metabolic Equivalent of Tasks (METs) and workload would indicate, it could be interpreted as a result of a higher glycogen formation leading to increased work output due to muscle signaling (Rauch et al, 2005). The current trial will allow 3 hours of absorption to estimate the likely benefit of phosphorus supplementation through enhanced glucose uptake possibly limited by phosphorus depletion under normal conditions, as noticed in the experiment of Khattab et al. (2015). The risk of change in blood osmolality due to administration of 100gr of Dextrose usually used in OGTT is minimal (Finta et al, 1992) .

Methods:

Inclusion criteria: AUB water polo players who are between the age of 18 and 25 years old, shall be included in the study.

Risk assessment: It should be noted that the university requires a clearance from Family Medicine following a general health and cardiac screening (ECG) for inclusion on a varsity team, which indicates that the trial includes no increased risk for the participating athletes. The health survey filled by the Family Medicine department physician includes presence of allergies and previous medical conditions.

A cross over study will be conducted on 17 male athletes (all members of the American University of Beirut's Water Polo Varsity Team), that are known to have similar energy expenditure and exercise patterns. Overnight fasted subjects will be depleted of glycogen. Participants will be asked to cycle for 20 min at 65% of each one's VO2max (that is determined prior to the experiment), thereafter will be given a meal (100g of glucose dissolved in 300 ml) with 4 tablets of phosphorus (100mg/tablet) or placebo in a random order.

Three hours later, participants will be asked to cycle for 40 mins, using the nutrition lab's CPET cyclometer and cardiopulmonary exercise testing machine COSMED at 80% their maximal heartrate (measured during a water polo training session). The heartrate during the training will be determined by using a waterproof heartrate monitor, PoolMateHR made by Swimovate and consisting of a specially designed low frequency detector that will transmit in water as explained by the makers. Body fat will be determined using the In-Body Bio-Electric Impedance machine at the nutrition lab. The ergometer will determine the METs and allow us to detect any potential ergogenic gain.

Procedure:

1. Identification and recruitment of subjects: Subjects will be approached at the swimming pool where the water polo training takes place. An overall briefing of the study will be given to the varsity players and if they are interested, then a detailed explanation will be given.
2. After reading and signing the consent form by both parties, participating athletes will be asked during their training session to wear a heartrate monitor, PoolMateHR made by Swimovate, to determine the heartbeat range during a typical training session which includes warm-up, drills and a water polo game.
3. On the day of the experiment following an overnight fast, the participant will be taken to the testing facility [Faculty of Agriculture and Food Sciences/Department of Nutrition and Food Science] where: anthropometric measurements will be taken (height, weight, WC), in addition to a body composition analysis using bioelectrical impedance analysis (BIA) where the individual will stand on a digital scale which runs an electrical current through the body in order to determine its composition (bones, fat, muscles, water, and their specific distributions)
4. The participant will be asked to cycle on the ergometer for 20 minutes at an average of 65% of the maximal heartrate that is determined during training, wearing the mouthpiece, to be familiar with the process. Afterwards, they will be served a flavored drink containing 100 g of glucose dissolved in 300 ml of water, with either 4 pills each containing 100 mg (total 400 mg) of phosphorus or placebo.
5. The participant will be asked to sit in a relaxed position and not to perform any major physical activity. Three hours later, he will be asked to cycle on the ergometer for 40 minutes at an average of 80% of the determined maximal heartrate during training while wearing the breathing mask.
6. The METs and workload will be measured using the CPET.

Analysis of Results:

Statistical Method:

Sample size was determined using the formula for two paired samples: n ≥ (σd /δd)2 (Zα+Zβ)2 which is reversely correlated to size effect, and directly correlated to Power. Since supplementation is relatively safe, especially at the low doses we use, and because any improvement is valuable, we opted for a Power between 70 and 80%.

Time trial results will compare workload and METs of two samples using a t-test, to estimate the effect of acute phosphate supplementation on glycogen replenishment. The hypothesized increase in workload after phosphate supplementation will be interpreted as the result of glycogen signaling leading to higher output as per the suggestion of glycogen signaling experiment (Rauch et al., 2005).

ELIGIBILITY:
Inclusion Criteria:

* water polo player

Exclusion Criteria:

-

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 17 (Estimated)
Dates: Start 2017-03-24 (Actual); Primary Completion 2018-03-24 (Estimated); Study Completion 2018-03-24 (Estimated)

PRIMARY OUTCOMES:
workload or performance enhancement or METs | up to 40 min
  power (watt) and time to exhaustion

CONTACTS AND LOCATIONS:
Overall Officials: omar obeid, PhD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buck CL, Wallman KE, Dawson B, Guelfi KJ. Sodium phosphate as an ergogenic aid. Sports Med. 2013 Jun;43(6):425-35. doi: 10.1007/s40279-013-0042-0. PMID 23568374
- [Background] Chasiotis D. Role of cyclic AMP and inorganic phosphate in the regulation of muscle glycogenolysis during exercise. Med Sci Sports Exerc. 1988 Dec;20(6):545-50. PMID 2853269
- [Background] Czuba M, Zajac A, Poprzecki S, Cholewa J, Woska S. Effects of Sodium Phosphate Loading on Aerobic Power and Capacity in off Road Cyclists. J Sports Sci Med. 2009 Dec 1;8(4):591-9. eCollection 2009. PMID 24149601
- [Background] Di Caprio G, Stokes C, Higgins JM, Schonbrun E. Single-cell measurement of red blood cell oxygen affinity. Proc Natl Acad Sci U S A. 2015 Aug 11;112(32):9984-9. doi: 10.1073/pnas.1509252112. Epub 2015 Jul 27. PMID 26216973
- [Background] Finta KM, Rocchini AP, Moorehead C, Key J, Katch V. Urine sodium excretion in response to an oral glucose tolerance test in obese and nonobese adolescents. Pediatrics. 1992 Sep;90(3):442-6. PMID 1518704
- [Background] Folland JP, Stern R, Brickley G. Sodium phosphate loading improves laboratory cycling time-trial performance in trained cyclists. J Sci Med Sport. 2008 Sep;11(5):464-8. doi: 10.1016/j.jsams.2007.04.004. Epub 2007 Jun 14. PMID 17569583
- [Background] Galloway SD, Tremblay MS, Sexsmith JR, Roberts CJ. The effects of acute phosphate supplementation in subjects of different aerobic fitness levels. Eur J Appl Physiol Occup Physiol. 1996;72(3):224-30. doi: 10.1007/BF00838643. PMID 8820890
- [Background] Khattab M, Abi-Rashed C, Ghattas H, Hlais S, Obeid O. Phosphorus ingestion improves oral glucose tolerance of healthy male subjects: a crossover experiment. Nutr J. 2015 Oct 29;14:112. doi: 10.1186/s12937-015-0101-5. PMID 26514124
- [Background] Kopec BJ, Dawson BT, Buck C, Wallman KE. Effects of sodium phosphate and caffeine ingestion on repeated-sprint ability in male athletes. J Sci Med Sport. 2016 Mar;19(3):272-276. doi: 10.1016/j.jsams.2015.04.001. Epub 2015 Apr 24. PMID 25953613
- [Background] Lichtman MA, Miller DR, Cohen J, Waterhouse C. Reduced red cell glycolysis, 2, 3-diphosphoglycerate and adenosine triphosphate concentration, and increased hemoglobin-oxygen affinity caused by hypophosphatemia. Ann Intern Med. 1971 Apr;74(4):562-8. doi: 10.7326/0003-4819-74-4-562. No abstract available. PMID 4994546
- [Background] Rauch HG, St Clair Gibson A, Lambert EV, Noakes TD. A signalling role for muscle glycogen in the regulation of pace during prolonged exercise. Br J Sports Med. 2005 Jan;39(1):34-8. doi: 10.1136/bjsm.2003.010645. PMID 15618337
- [Background] Xie W, Tran TL, Finegood DT, van de Werve G. Dietary P(i) deprivation in rats affects liver cAMP, glycogen, key steps of gluconeogenesis and glucose production. Biochem J. 2000 Nov 15;352 Pt 1(Pt 1):227-32. PMID 11062077
- [Derived] Elhusseini R, Fares EJ, Obeid O. Phosphorus supplementation raised the heart rate of male water polo players during a randomised graded dryland exercise test. BMJ Open Sport Exerc Med. 2020 Apr 8;6(1):e000714. doi: 10.1136/bmjsem-2019-000714. eCollection 2020. PMID 32405431